CLINICAL TRIAL: NCT00843154
Title: Effects Of Candesartan Cilexetil vs Standard Therapy on Serum Levels of Brain Natriuretic Peptide in Patients Suffering From Chronic Heart Failure With Depressed and Preserved Systolic Function
Brief Title: Efficacy of Candesartan on Brain Natriuretic Peptide Levels in Subjects With Chronic Heart Failure
Acronym: CANDHEART
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Italia Farmaceutici SpA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CANc-CHF14-TIF; 2005-001306-87 (EudraCT Number); U1111-1114-0042 (Registry Identifier: WHO)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Heart Failure
Keywords: Natriuretic Peptide, Brain; Biological Markers; Biomarkers; Cardiac Failure; Congestive Heart Failure; Heart Decompensation; Drug Therapy
MeSH Terms: conditions — Heart Failure | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan QD (Experimental)
  Interventions: Drug: Candesartan and standard chronic heart disease therapy
- Standard chronic heart disease therapy (Active Comparator)
  Interventions: Drug: Standard chronic heart disease therapy

INTERVENTIONS:
Drug: Candesartan and standard chronic heart disease therapy — Candesartan 4mg, tablets, orally, once daily and stable dose therapy for chronic heart disease for two weeks; then Candesartan increased up to 32mg, tablets, orally, once daily and stable dose therapy for chronic heart disease for up to 48 weeks.
  Other Names: Blopress; Amias; Kenzen; Atacand; Blopressid
  Arms: Candesartan QD
Drug: Standard chronic heart disease therapy — Candesartan placebo-matching tablets, orally, once daily and stable dose therapy for chronic heart disease for up to 48 weeks.
  Arms: Standard chronic heart disease therapy

SUMMARY:
The purpose of this study is to determine the effects of Candesartan, once daily (QD), added to ongoing chronic heart disease therapy in measuring brain natriuretic peptide in patients with chronic heart failure.

DETAILED DESCRIPTION:
Chronic heart failure is a significant and increasing cause of morbidity and mortality, accounting for a current yearly prevalence of 5 million and a 5-year survival near 50% in the US. In addition, chronic heart failure is still the fourth cause of hospitalization in the US and in Western countries, and it is the leading cause of hospitalization in patients aged over 65.

Newer pharmacological agents and non pharmacological therapeutic tools have been increasingly introduced to improve the outcomes in patients with chronic heart failure. In the past two decades, several large randomized controlled clinical trials have revolutionized the management and prognosis of patients with chronic heart failure. The recommended drug treatment for decreasing mortality and morbidity in chronic heart failure is based on angiotensin converting enzyme-inhibitors, beta-blockers and aldosterone antagonists (limited to most severe patients), as detailed in the latest European Society of Cardiology guidelines. The use of digitalis and diuretics still has a role.

Orally active angiotensin II type I receptor blockers represent a new class of agents that offer an alternative method of the renin-angiotensin system blockade. Their effects on hemodynamics, neuroendocrine activity and exercise tolerance in patients with chronic heart failure can be considered as similar to that exhibited by angiotensin converting enzyme -inhibitors, but it still remains to be fully elucidated whether angiotensin II type I receptor blockers can offer advantage in efficacy, other than in safety, compared to angiotensin converting enzyme -inhibitors.

Brain Natriuretic Peptide is strongly related to the severity and to the increase of cardiovascular events in patients with chronic heart failure. Recent data show that angiotensin II receptor blockers can reduce the levels of Brain Natriuretic Peptide, though no data is available in patients with preserved left ventricular systolic function.

Candesartan is a selective angiotensin II type I receptor blocker, and this study will evaluate the effects of the maximum tolerated dose of Candesartan added to ongoing standard therapy while measuring changes in brain natriuretic peptide biomarker used in the assessment of chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Stable, symptomatic New York Heart Association II-IV Chronic Heart Failure with Left Ventricular Ejection Fraction less than or greater than or greater than or equal to 40% treated with standard therapy including Angiotensin Converting Enzyme-inhibitors and/or beta-blockers. Patients with Left Ventricular Ejection Fraction greater than or equal to 40% had to be hospitalized for cardiovascular events during the past 12 months.

Exclusion Criteria:

* History of prior treatment with Angiotensin-Receptor Blockers within two weeks from first.
* Severe or malignant hypertension (Systolic Blood Pressure / Diastolic Blood Pressure greater than 180/110 mmHg).
* Symptomatic hypotension.
* Acute myocardial infarction within one month from first visit.
* Stroke or transient ischemic attack within one month from first visit.
* Percutaneous transluminal coronary angioplasty or coronary artery by-pass graft within one month from first visit.
* Hemodynamically relevant arrhythmias.
* Implant of pacemakers, cardiac resynchronization therapy or cardioverters within 6 months prior the randomization.
* Hemodynamically relevant cardiac valvular defect.
* Constrictive pericarditis or active myocarditis.
* Likelihood of cardiac surgical intervention (of any type) during the overall treatment period.
* Evidence of angina pectoris in the previous month.
* Poorly controlled diabetes mellitus (glycemia greater than 140mg/mL or glycosylated hemoglobin greater than 8% obtained within three months from the study initiation).
* Untreated thyroid dysfunction.
* Renal artery stenosis.
* Angioedema of any etiology.
* Significant liver (aspartate aminotransferase, alanine aminotransferase, total bilirubin or alkaline phosphatase greater than twice the upper limit of normal range) or renal (serum creatinine greater than 2.0 mg/dL or serum potassium greater than 5.0 mmol/L) impairment.
* Anemia of any etiology (defined as hemoglobin levels less than 10.5 g/dL) or any other clinically relevant hematological disease.
* Any disease with malabsorption.
* Presence of any non-cardiac (e.g. cancer) disease that is likely to significantly (i.e. below 1 year from randomization) shorten life expectancy.
* History of chronic alcohol or drug/substance abuse, or presence of other conditions potentially able to affect study subjects' compliance.
* Known allergy, sensitivity or intolerance to study drugs and/or study drugs' formulation ingredients.
* Participation in another trial in the month preceding study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2005-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Brain Natriuretic Peptide | Week 12 or Final Visit.

SECONDARY OUTCOMES:
Change from baseline in Brain Natriuretic Peptide | Week 48 or Final Visit.
Change from baseline in Aldosterone, Pentraxin-3 and C-Reactive Protein | Week 48 or Final Visit.
Change from baseline of New York Heart Association class | Week 48 or Final Visit.
Change from baseline of Left Ventricular Ejection Fraction, Left Ventricular Internal Diastolic Diameter, E wave peak velocity/A wave peak velocity, deceleration time of E wave, atrial dimensions, blood pressure and heart rate | Week 48 or Final Visit.
Persistence of active treatment and discontinuation rate | Week 48 or Final Visit.
Quality of life as measured by Kansas City Cardiomyopathy Questionnaire | Week 48 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Director, Study Director — Takeda Italia Farmaceutici SpA